CLINICAL TRIAL: NCT01096771
Title: The Effect of Intravenous Lipid Emulsions on Lung Function in ARDS: A Pilot Study
Brief Title: The Effect of Intravenous Lipids on Lung Function in Acute Respiratory Distress Syndrome (ARDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to secure product from international source, low recruitment rate.
Sponsor: Methodist Research Institute, Indianapolis (Other)
Responsible Party: Principal Investigator, W. Graham Carlos, MD, Methodist Research Institute, Indianapolis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Lipids for ARDS
Record Dates: First submitted 2010-03-24; First posted 2010-03-31 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Parenteral; Pharmaconutrition
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ClinOleic 20% (Experimental): 96 hour continuous infusion.
  Interventions: Drug: ClinOleic 20%
- Intralipid 20% (Active Comparator): 96 hour continuous infusion.
  Interventions: Drug: Intralipid 20%

INTERVENTIONS:
Drug: ClinOleic 20% — 96 hour continuous infusion.
  Arms: ClinOleic 20%
Drug: Intralipid 20% — 96 hour continuous infusion.
  Arms: Intralipid 20%

SUMMARY:
The purpose of this study is to evaluate the effects of nutritional supplementation with omega-9 "olive-oil" and omega-6 "soybean oil" based lipid emulsions in the Acute Respiratory Distress Syndrome (ARDS). The investigators hypothesize that these specific lipids in combination will immunomodulate the inflammatory reaction that occurs in the lungs of ARDS subjects. This concept is known as "Pharmaconutrition." These lipids will be given intravenously so as to assure administration and only as a supplement to enteral nutrition which all subjects will also receive. The omega-9 will be compared to the omega-6 formulation which is the only FDA approved formulation of use in the United States since its development in 1961 by Fresenius-Kabi, Bad Homburg, Germany. The investigators plan to perform a bronchoscopy with lavage within 24 hours of enrollment, begin the lipid administration and continue it for 96 hours after which time the investigators will repeat bronchoscopy with lavage to assess changes. The lipid administration will cease following the second bronchoscopy. The fluid obtained from lavage combined with serum samples obtained at the time of bronchoscopy will be analyzed for inflammatory mediators and cell counts. Clinical data tracing will include but not be limited to: ventilator days, nutritional status, ICU time, oxygenation and lung compliance, and 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with predisposing condition causing ARDS
* are mechanically ventilated through an endotracheal tube
* have enteral feeding access
* have central venous access
* have a PaO2:FiO2 ratio of less than 200
* have bilateral pulmonary infiltrates on chest x-ray

Exclusion Criteria:

* sedation requiring the use of diprivan (after enrollment)
* a clinical diagnosis of left ventricular failure
* lung cancer
* hematologic malignancy
* severe dyslipidemia
* condition precluding bronchoscopy including inability to maintain oxygen saturations greater than 90% per pulse oximetry despite conventional mechanical ventilation
* severe immunosuppression
* use of NSAIDS within previous 24 hours
* HIV positive
* pregnancy
* hypersensitivity to egg or soybean oil
* active myocardial infarction
* acute pancreatitis if complicated by hypertriglyceridemia
* severe sepsis with 2 or more organ failures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Naum, MD, Principal Investigator — Indiana Clinic
Locations (1):
- Methodist Hospital, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental ClinOleic 20%: Patients received dietary supplement with ClinOleic 20%.
- Control: Intralipid 20%: Patients received dietary supplement with Intralipid 20%.
Period: Overall Study
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20% | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11.24) | 60 (14.55) | 62 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Bronchoalveolar Lavage Fluid Interleukin-8 Concentrations
Time Frame: 96 hours
Population: Each arm has one less subject than specified in the participate flow module. One is secondary to the fact that the subject refused the 2nd bronchoscopy and the other is because the primary physician felt the subject was too sick to undergo the 2nd bronchscopy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Number analyzed (Participants) | 6 | 6
pg/mL | 1092 (1017) | 544 (453.6)

2. Secondary Outcome: Ventilator Days
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Number analyzed (Participants) | 7 | 7
days | 18 (10.11) | 18 (11.34)

3. Secondary Outcome: PaO2:FiO2 Ratio
Description: PaO2:FiO2 ratio at time of 2nd Bronchoalveolar Lavage (BAL) or end of study drug administration.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Number analyzed (Participants) | 7 | 7
mmHg | 159 (60.8) | 149 (78.44)

4. Secondary Outcome: 30 Day Mortality
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Number analyzed (Participants) | 7 | 7
participants | 1 | 1

5. Secondary Outcome: New Infection
Description: We will use standard clinical criteria including but not limited to: fever, pyuria, new inflitrate on chest x-ray, positive blood cultures, abscess detected on imaging, leukocytosis, and positive skin or soft-tissue cultures to identify presence of new bacterial infections occurring after enrollment.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Number analyzed (Participants) | 7 | 7
participants | 1 | 0

6. Secondary Outcome: Organ Failures
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Number analyzed (Participants) | 7 | 7
participants | 1 | 1

7. Secondary Outcome: Biomarkers (C-reactive Protein)
Time Frame: 96 hours
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Number analyzed (Participants) | 7 | 7
mg/L | 10 (9.06) | 13 (13.81)

8. Secondary Outcome: Hospital Length of Stay
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Number analyzed (Participants) | 7 | 7
days | 22 (8.45) | 28 (19.78)

9. Secondary Outcome: Allergic Reactions
Time Frame: 96 hours
Measure: Number; unit: participants
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Number analyzed (Participants) | 7 | 7
participants | 0 | 0

10. Secondary Outcome: Hypertriglyceridemia
Description: Defined as triglyceride level >400
Time Frame: 96 hours
Measure: Number; unit: participants
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Number analyzed (Participants) | 7 | 7
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Experimental ClinOleic 20% | Control: Intralipid 20%
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/7
Other Adverse Events (participants affected / at risk) | 1/7 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental ClinOleic 20% (N=7) | Control: Intralipid 20% (N=7)
Death (Cardiac disorders) | 1 (1) | 1 (1) — Patient died after study infusion drug completed. Mortality rate for ARDS is >25%. While this is a SAE it is not unexpected and could not be directly connected to study experimental or control drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental ClinOleic 20% (N=7) | Control: Intralipid 20% (N=7)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1) — An adverse event was considered a rise in the serum creatinine level while on the study experimental or control drug.
New Infection (Infections and infestations) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No